CLINICAL TRIAL: NCT07288424
Title: Implementation and Efficacy of an Opioid-Free Analgesic Regimen for Postoperative Pain Management in Adolescent Patients With Pectus Excavatum After NUSS Surgery
Brief Title: Opioid-Free Pain Management After NUSS Surgery in Adolescents
Status: Completed | Type: Observational
Sponsor: Qin Zhang (Other)
Responsible Party: Sponsor-Investigator, Qin Zhang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Other Study IDs: TJ-IRB202509077
Record Dates: First submitted 2025-11-23; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Nerve Block
Keywords: Nerve Block
MeSH Terms: interventions — Nerve Block

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: Patients who underwent ultrasound-guided bilateral transverse thoracic fascia block and intercostal nerve block after general anesthesia induction but before surgery.
  Interventions: Procedure: Nerve block
- Control group: Patients who received incision local infiltration, serratus anterior plane block, intercostal nerve block, and erector spinae plane block.

INTERVENTIONS:
Procedure: Nerve block — Ultrasound-guided bilateral transverse thoracic fascia block and intercostal nerve block
  Groups: Experimental group

SUMMARY:
The investigators applied ultrasound-guided bilateral transverse thoracic fascia block combined with intercostal nerve block-a previously unreported analgesic approach for post-thoracic surgery-to NUSS patients. These suggest that ultrasound-guided transverse thoracic fascia combined with intercostal nerve block, in conjunction with bupivacaine liposome (72-hour analgesic duration), holds promise for a clinically feasible opioid-free analgesic regimen for severe post-NUSS pain.

DETAILED DESCRIPTION:
Performance of Nerve Blocks and Data collection Transverse thoracic fascia block: Under ultrasound guidance, the deep layer of the transverse thoracic fascia was localized at the parasternal 4th-5th intercostal space, with 10 mL of local anesthetic mixture (bupivacaine liposome 4mg/kg + 0.75% bupivacaine injection 5mL, diluted to 32mL with normal saline) injected on each side.

Intercostal nerve block: The 4th-8th intercostal spaces were identified at the posterior axillary line level. Under ultrasound guidance, the local anesthetic was injected between the internal intercostal and innermost intercostal muscles, with 2 mL of the aforementioned mixture administered per intercostal space.

Multimodal Analgesia Regimen

First, 50 mg of flurbiprofen axetil injection was intravenously administered before the surgeon made the skin incision. Second, 0.07 mg/kg of oxycodone was intravenously injected 30 minutes before the end of surgery. Third, a patient-controlled intravenous analgesia (PCA) pump was connected upon admission to the Post-Anesthesia Care Unit (PACU). After transfer to the ward, if the patient's pain score was ≥ 4 points, ward doctors administered diclofenac sodium via anal suppository.

Pain Assessment and Management Measures

Pain was assessed every 2 hours within 12 hours postoperatively (upon admission to the PACU, 2 hours, 4 hours, 6 hours, and 12 hours postoperatively) and every 4 hours from 12 to 72 hours postoperatively. Pain scores were recorded at each time point using a Visual Analogue Scale (VAS). Additionally, the time and dose of supplementary analgesics administered were documented, and pain relief efficacy was reassessed and recorded 2 hours after administration.

Study Population

This study enrolled children and adolescents who underwent the NUSS procedure for pectus excavatum at the Department of Thoracic Surgery, Tongji Hospital, from June to September 2025. The inclusion criterion was age between 8 and 18 years (inclusive). Patients who received epidural analgesia or bilateral paravertebral nerve blocks were excluded.

Experimental group: Patients who underwent ultrasound-guided bilateral transverse thoracic fascia block and intercostal nerve block after general anesthesia induction but before surgery.

Control group: Patients who received incision local infiltration, serratus anterior plane block, intercostal nerve block, and erector spinae plane block.

Study Variables The investigators collected relevant variables based on the quality of postoperative recovery in NUSS patients reported in the literature. Data Collection and Measurement of Variables: Demographic data of patients were collected upon hospital admission. Pain was assessed using a Visual Analogue Scale (VAS).Time and dose of additional postoperative analgesic drugs; Postoperative recovery indicators: breathing pain, compulsive posture, postoperative hospital stay, oxygen inhalation rate exceeding 24 hours after operation.

Statistical Analysis R studio was used for statistical analysis in this study. Categorical data were expressed as counts (percentages) [n(%)], and comparisons between groups were performed using the chi-square test; if the theoretical frequency was <5, Fisher's exact test was applied. Normality test was first performed for continuous data. Continuous data conforming to normal distribution were presented as mean ± standard deviation (x±s), and independent samples t-test was used for intergroup comparisons, while repeated measures analysis of variance (ANOVA) was used for intragroup comparisons at different time points. Continuous data not conforming to normal distribution were expressed as median (interquartile range) [M(Q1,Q3)], and intergroup comparisons were conducted using the Mann-Whitney U test. A P value <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents who underwent the NUSS procedure.
* Adolescents who were between 8 and 18 years .

Exclusion Criteria:

* Adolescents who received epidural analgesia.
* Adolescents who received bilateral paravertebral nerve blocks.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study enrolled children and adolescents who underwent the NUSS procedure for pectus excavatum at the Department of Thoracic Surgery, Tongji Hospital, from June to September 2025. The inclusion criterion was age between 8 and 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Pain score | 72 hours
  Pain was assessed every 2 hours within 12 hours postoperatively (upon admission to the PACU, 2 hours, 4 hours, 6 hours, and 12 hours postoperatively) and every 4 hours from 12 to 72 hours postoperatively. Pain scores were recorded at each time point using a Visual Analogue Scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Qin Zhang, phd, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No